CLINICAL TRIAL: NCT05375669
Title: The Effect of Increasing Current or Pulse Duration on Patient Movement and Intraoperative Transcranial Electric Stimulation Motor Evoked Potential Amplitude
Acronym: CCCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCV
Record Dates: First submitted 2022-04-21; First posted 2022-05-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: Patients will be screened as part of the clinical routine and will be included if they satisfy the eligibility criteria and sign the informed consent. All the study subjects who are included are patients who undergo surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ISIS IOM System (Experimental): Total intravenous anesthesia (TIVA), surgery and TES MEP monitoring will proceed routinely without modification and normally involves acquiring many MEPs over several hours. The only departure from standard care will be the placement of two small accelerometers and a brief MEP sequence before skin incision to determine chronaxie and compare the effect of an equivalent increase of I or D on MEP amplitude and movement.
  Interventions: Device: ISIS IOM System

INTERVENTIONS:
Device: ISIS IOM System — The constant-current TES stimulators will be used in this study with a high-precision oscilloscope. The calibration will assess 5-pulse trains with a 4 ms ISI and 100 mA output across a 1000 Ω resistor at 250, 500, and 1000 µs D. Measurements will include actual I and D of each pulse, and actual ISI.
  Total intravenous anesthesia (TIVA), surgery and TES MEP monitoring will proceed routinely without modification and normally involves acquiring many MEPs over several hours. The only departure from standard care will be the placement of two small accelerometers and a brief MEP sequence before skin incision to determine chronaxie and compare the effect of an equivalent increase of I or D on MEP amplitude and movement.

SUMMARY:
Transcranial electric stimulation (TES) motor evoked potential (MEP) monitoring is standard during surgery risking motor system injury. The stimuli are typically 5-pulse trains with a 4 ms interstimulus interval (ISI). The pulse duration (D) is often set to 50 or 500 µs. Both are effective, but setting D to the chronaxie would be physiologically optimal and limited data suggest that mean MEP chronaxie may be near 200 µs.

When necessary, one can obtain larger MEPs by increasing current (I) or D to increase stimulus charge (Q = I × D). However, this also increases patient movement that can interfere with surgery and reduce MEP acquisition frequency.

The main research question is whether increasing current or pulse duration when applying intraoperative neuromonitoring produces less patient movement during surgery. As such, the IOM ISIS System will be employed for neuromonitoring and an accelerometer will be used to quantify patient movement.

The constant-current TES stimulators will be used in this study with a high-precision oscilloscope. Total intravenous anesthesia (TIVA), surgery and TES MEP monitoring will proceed routinely without modification and normally involves acquiring many MEPs over several hours. The only departure from standard care will be the placement of two small accelerometers and a brief MEP sequence before skin incision to determine chronaxie and compare the effect of an equivalent increase of I or D on MEP amplitude and movement.

DETAILED DESCRIPTION:
Transcranial electric stimulation (TES) motor evoked potential (MEP) monitoring is standard during surgery risking motor system injury. The stimuli are typically 5-pulse trains with a 4 ms interstimulus interval (ISI). The pulse duration (D) is often set to 50 or 500 µs. Both are effective, but setting D to the chronaxie would be physiologically optimal and limited data suggest that mean MEP chronaxie may be near 200 µs.

When necessary, one can obtain larger MEPs by increasing current (I) or D to increase stimulus charge (Q = I × D). However, this also increases patient movement that can interfere with surgery and reduce MEP acquisition frequency. Anecdotal observations suggest that increasing D may produce larger MEPs with less movement than increasing I, but there is no published support. If true, then the optimal D for monitoring may be above the chronaxie because less movement could facilitate more frequent MEP acquisition.

Finally, there is ongoing controversy about constant-current or constant-voltage TES. However, with stable resistance (R) there is no fundamental reason to prefer one or the other since they are related by Ohm's law I = V/R. Also, since threshold current and voltage vary with D their maximum levels should also vary with selected D, which could be confusing. Instead, because the International Electrotechnical Commission 50 mJ safety limit is based on energy (E = I2 × D × R = V2 × D/R), it may be more logical to apply constant-energy TES that would provide a consistent 0-50 mJ selection range at any selected D.

The primary objective is to assess whether intraoperative neuromonitoring with constant current or constant voltage produces less patient movement during surgery. The secondary objectives are to compare MEP amplitudes with the different setups, to estimate the true mean or median chronaxie and to develop the concept of constant-energy TES.

The main research question is whether increasing current or pulse duration when applying intraoperative neuromonitoring produces less patient movement during surgery. As such, the IOM ISIS System will be employed for neuromonitoring and an accelerometer will be used to quantify patient movement.

The constant-current TES stimulators will be used in this study with a high-precision oscilloscope. The calibration will assess 5-pulse trains with a 4 ms ISI and 100 mA output across a 1000 Ω resistor at 250, 500, and 1000 µs D. Measurements will include actual I and D of each pulse, and actual ISI.

Total intravenous anesthesia (TIVA), surgery and TES MEP monitoring will proceed routinely without modification and normally involves acquiring many MEPs over several hours. The only departure from standard care will be the placement of two small accelerometers and a brief MEP sequence before skin incision to determine chronaxie and compare the effect of an equivalent increase of I or D on MEP amplitude and movement.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* The patient has a supra- or infra-tentorial lesion requiring surgery
* The patient is undergoing neurosurgery with the use of Intraoperative Monitoring (IOM) during surgery to protect functional tissue
* The patient is older than 18 years

Exclusion Criteria:

* No need for Intraoperative Monitoring (IOM)
* Vulnerable subjects (pregnant women, pregnant, impaired consciousness)
* People who do not want to participate in the study
* Emergency procedures in which no consent was obtained before the operation
* Multiple surgeries on the same patient
* Preoperative non-affected arm motor deficit (MRC <5), that is to say, no motor deficit of the arm ipsilateral to the surgery
* Inhalational anesthesia
* Persisting neuromuscular blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of a 2-fold increase of I or of D from threshold on patient movement | During surgery, estimated on average to be about 4 hours
  Comparison of the effect of a 2-fold increase of I or of D from threshold on patient movement quantified by accelerometers on the patient's forehead and contralateral (non-affected) shoulder.

SECONDARY OUTCOMES:
Comparing the effect of a 2-fold increase of I or of D from threshold on MEP amplitude | During surgery, estimated on average to be about 4 hours
  Compare the effect of a 2-fold increase of I or of D from threshold on MEP amplitude as measured by the ISIS IOM System
Chronaxie | During surgery, estimated on average to be about 4 hours
  The stimulation strength (in mA) necessary to elicit an MEP are measured with the different pulse durations (in μs)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Seidel, MMD, Principal Investigator — Inselspital Bern, Department of Neurosurgery
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szelenyi A, Kothbauer KF, Deletis V. Transcranial electric stimulation for intraoperative motor evoked potential monitoring: Stimulation parameters and electrode montages. Clin Neurophysiol. 2007 Jul;118(7):1586-95. doi: 10.1016/j.clinph.2007.04.008. Epub 2007 May 15. PMID 17507288
- [Background] Abalkhail TM, MacDonald DB, AlThubaiti I, AlOtaibi FA, Stigsby B, Mokeem AA, AlHamoud IA, Hassounah MI, Baz SM, AlSemari A, AlDhalaan HM, Khan S. Intraoperative direct cortical stimulation motor evoked potentials: Stimulus parameter recommendations based on rheobase and chronaxie. Clin Neurophysiol. 2017 Nov;128(11):2300-2308. doi: 10.1016/j.clinph.2017.09.005. Epub 2017 Sep 28. PMID 29035822
- [Background] Macdonald DB, Skinner S, Shils J, Yingling C; American Society of Neurophysiological Monitoring. Intraoperative motor evoked potential monitoring - a position statement by the American Society of Neurophysiological Monitoring. Clin Neurophysiol. 2013 Dec;124(12):2291-316. doi: 10.1016/j.clinph.2013.07.025. Epub 2013 Sep 18. PMID 24055297
- [Background] MacDonald DB. Safety of intraoperative transcranial electrical stimulation motor evoked potential monitoring. J Clin Neurophysiol. 2002 Oct;19(5):416-29. doi: 10.1097/00004691-200210000-00005. PMID 12477987
- [Background] Eng J. Sample size estimation: how many individuals should be studied? Radiology. 2003 May;227(2):309-13. doi: 10.1148/radiol.2272012051. PMID 12732691